CLINICAL TRIAL: NCT07092553
Title: Evaluation of C-arm Photon Counting Detector Cone Beam CT (PCD-CBCT) for Image-Guided Interventions
Brief Title: Evaluation of C-arm PCD-CBCT for Image-Guided Interventions
Status: Not yet recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2025-0677; 1R01EB034011-01A1 (NIH); A534800 (Other: UW Madison); SMPH/MED PHYSICS/MED PHYSIC (Other: UW Madison); Protocol Version 3/10/2025 (Other: UW Madison)
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-07

CONDITIONS: Imaging
Keywords: image-guided intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients with SOC image-guided intervention: Patients undergoing a standard of care (SOC) image-guided intervention of the head or body
  Interventions: Device: C-arm PCD-CBCT

INTERVENTIONS:
Device: C-arm PCD-CBCT — A single research PCD-CBCT scan will be performed directly after the participant's SOC scan.

SUMMARY:
The overarching objective of the project is to develop a new C-arm interventional x-ray imaging platform that integrates both a photon counting detector and a flat panel detector to provide high image quality and quantitative spectral computed tomography (CT) image guidance will be developed to enable more accurate and safe interventional procedures for patients.

DETAILED DESCRIPTION:
The objective of this pilot study is to assess the feasibility of acquiring high-quality images using new imaging concepts and methods. All imaging will be performed in addition to standard-of-care procedures and will not influence clinical decisions or patient management.

The endpoint of this project includes: 1) PCD-CBCT data will be processed to generate virtual non-iodine images for evaluating contrast extravasation, as well as virtual monoenergetic (VME) images. 2) Images will be analyzed retrospectively to evaluate image quality and explore potential clinical benefits of PCD-CBCT compared to flat panel detector cone beam CT (FPD-CBCT) and multidetector computed tomography (MDCT).

ELIGIBILITY:
Inclusion Criteria:

* Not pregnant or breastfeeding
* Scheduled to receive image-guided intervention (IGI) of the head or the body
* Pre-treatment multidetector computed tomography (MDCT) images available

Exclusion Criteria:

* Unable to provide informed consent on their own behalf due to cognitive impairment
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a SOC image-guided intervention of the head or body
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Mean Confidence Score for Calcifications | after participant data collection is complete (up to 1 year)
  MDCT, PCD-CBCT, and FPD-CBCT images will be co-registered and displayed on a clinical monitor using a customized software that allows the users to toggle between energy bin images. At least 4 readers with a broad spectrum of clinical experiences (radiology residents, interventional radiology and neurosurgery fellows, and experienced physician co-investigators) will independently identify calcifications and extravasated iodine contrast (if available) and provide a 1 (low) to 5 (high) confidence score on each image.
Mean Confidence Score for Metal Artifacts | after participant data collection is complete (up to 1 year)
  MDCT, PCD-CBCT, and FPD-CBCT images will be co-registered and displayed on a clinical monitor using a customized software that allows the users to toggle between energy bin images. At least 4 readers with a broad spectrum of clinical experiences (radiology residents, interventional radiology and neurosurgery fellows, and experienced physician co-investigators) will independently identify metal artifacts (if any) and provide a 1 (low) to 5 (high) confidence score on each image.
Area Under the Curve (AUC) for Calcification Detection | image analysis will proceed after participant data collection is complete (up to 2 years)
  For all reading studies, the order of subjects and imaging modality (MDCT, FPD-CBCT, and PCD-CBCT) will be randomized; three separate reading sessions will be implemented with a washout period of at least 3 months between sessions.
  For calcification and iodine staining detection in the human subjects, the receiver operating characteristic (ROC) curves will be calculated using the maximum-likelihood method with the binormal model. The 95% confidence interval (CI) of each ROC curve will be estimated and the area under the curve (AUC) and its 95% CI will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Guang-Hong Chen, PhD, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- UW Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No